CLINICAL TRIAL: NCT06429579
Title: Multicenter, Prospective, and Exploratory Study of Potts-shunt for the Treatment of Pediatric Patients With Severe Pulmonary Hypertension
Brief Title: Potts-shunt for the Treatment of Pediatric Patients With Severe Pulmonary Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCRC2024001
Record Dates: First submitted 2024-05-05; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potts-shunt combined with conventional drug therapy group (Experimental): The comprehensive therapy included Potts-shunt procedure and conventional drug therapy (i.e., Prostacyclin analogues, PDE-5 inhibitors, and Endothelin receptor antagonists)
  Interventions: Procedure: Comprehensive therapy combined Potts-shunt procedure and conventional drug therapy
- Only conventional drug therapy group (Active Comparator): Only admitted with conventional drug therapy (i.e., Prostacyclin analogues, PDE-5 inhibitors, and Endothelin receptor antagonists)
  Interventions: Drug: Only conventional drug therapy

INTERVENTIONS:
Procedure: Comprehensive therapy combined Potts-shunt procedure and conventional drug therapy — Potts-shunt procedure is the surgery that connect the descending aorta and the left/main pulmonary artery by direct anastomosis, a Gore-tex tube or a Gore-tex tube with flap.
  Arms: Potts-shunt combined with conventional drug therapy group
Drug: Only conventional drug therapy — Only conventional drug therapy (i.e., Prostacyclin analogues, PDE-5 inhibitors, and Endothelin receptor antagonists)
  Arms: Only conventional drug therapy group

SUMMARY:
This is a multi-center, perspective, and exploratory study aimed at evaluating the 3-years clinical outcome of Potts-shunt procedure for pediatric patients with severe pulmonary artery hypertension (PAH). The included criteria are as followed: 1)6 months < age ≤ 18 years; 2) ESC 2022 Group I PAH; 3) Have received standardized drug therapy for at least 6-9 months and still remain at intermediate to high/high-risk status of the criteria of ESC2022; 4) Presenting with significant clinical manifestations (i.e., progressive symptoms/syncope history/growth and development restriction, etc); 5) Informed consent form signed by the patient and their guardian. The excluded criteria are as followed: 1) ESC 2022 Group II-V PAH; 2) Poor right ventricular function: RVEF < 25% or RVFAC < 20%; 3) Deteriorated general condition: requiring ICU resuscitation or ECMO assistance; 4) Pulmonary artery pressure/main arterial pressure ratio < 0.7; 5) Six-minute walk distance < 150 meters (only applicable to patients aged 8 and above); 6) No significant improvement in RVEF under triple drug therapy. All of the pediatric patients with severe PAH who attend to pediatric cardiac outpatient clinic and meet the designed included criteria and excluded criteria will be enrolled in this study. All of the participants will be divided into two groups (Potts-shunt combined with conventional drug therapy group and only conventional drug therapy group) according to their individual health status (i.e., some contraindications of surgery) and their (or their parents') aspiration for Potts-shunts procedure. Follow-up is designed (eight-times follow-up) at the time of Potts-shunt procedure, post-operative ICU period, one month, three months, six months, one year, two years, and three years after Potts-shunt procedure or the rejection of Potts-shunt procedure. The items of follow-up include state of survival, whether or not have the lung transplantation (LTx), clinical manifestation, laboratory examination, function of right ventricle (detected by echocardiogram and cardiac magnetic resonance imaging), and the pulmonary circulation pressure (detected by right heart catheterization or Swan-Ganz catheterization). Primary outcome is the incidence rates of death or LTx three-years after Potts-shunt. Secondary outcomes are as followed: 1) Number and incidence rate of postoperative complications in patients undergoing Potts-shunt procedure; 2) Three-year WHO cardiac functional and 6-minute walk distance after Potts-shunt procedure; 3) the NT-ProBNP levels three-years after Potts-shunt procedure; 4) Right ventricular function on echocardiography three years after Potts-shunt procedure; 5) Right ventricular function on cardiac magnetic resonance imaging three years after Potts-shunt procedure; 6) Pulmonary circulation pressure measured by right heart catheterization or Swan-Ganz catheterization three years after Potts-shunt procedure; 7) Three-year mortality or LTx incidence rates after only conventional drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 6 months < age ≤ 18 years;
2. ESC 2022 Group I PAH;
3. Have received standardized drug therapy for at least 6-9 months and still remain at intermediate to high/high-risk status of the criteria of ESC2022;
4. Presenting with significant clinical manifestations (i.e., progressive symptoms/syncope history/growth and development restriction, etc);
5. Informed consent form signed by the patient and their guardian.

Exclusion Criteria:

1. ESC 2022 Group II-V PAH;
2. Poor right ventricular function: RVEF < 25% or RVFAC < 20%;
3. Deteriorated general condition: requiring ICU resuscitation or ECMO assistance;
4. Pulmonary artery pressure/main arterial pressure ratio < 0.7;
5. Six-minute walk distance < 150 meters (only applicable to patients aged 8 and above);
6. No significant improvement in RVEF under triple drug therapy.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2029-04-23 (Estimated); Study Completion 2029-04-23 (Estimated)

PRIMARY OUTCOMES:
Mortality or Lung transplantation | From the date of enrollment until the date of dear from any cause or lung transplantation, which ever came first, accessed up to 3 years
  The incidence rates of death or lung transplantation 3 years after Potts-shunt, accessed by in-patient, out-patient, or telephone follow-up

SECONDARY OUTCOMES:
Number and incidence rate of postoperative complications in patients undergoing Potts-shunt procedure | From the date of enrollment to the date of any postoperative complications, whichever came first, accessed up to 3 years
  Postoperative complications include hemoptysis, syncope, pulmonary hypertension crisis, low blood oxygen in the lower extremities etc. accessed by pediatric ICU doctors.
World Health Organization functional class (WHO-FC) after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  WHO-FC was designed to measure the severity of pulmonary hypertension based on symptoms of dyspnea, fatigue, chest pain, and related syncope, accessed by the pediatric doctors.
NT-ProBNP levels after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  NT-ProBNP (pg/ml) accessed by laboratory test
Right ventricular function on cardiac magnetic resonance imaging after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  The RVEF (%) accessed by cardiac MRI
Right ventricular function on echocardiography after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  The RVFAC (%) accessed by echocardiography
Pulmonary circulation pressure measured by right heart catheterization or Swan-Ganz catheterization after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  SPAP, DPAP, MPAP (mmHg) etc. accessed by right heart catheterization or Swan-Ganz catheterization
Mortality or lung transplantation incidence rates after only conventional drug therapy | From the date of enrollment until the date of dear from any cause or lung transplantation, which ever came first, accessed up to 3 years
  The incidence rates of death or lung transplantation 3 years after enrollment
The 6-minutes distance after Potts-shunt procedure | From the date of enrollment to the date of every view-point, assessed up to 3 years
  The 6-minutes distance (meter) was designed to measure activity tolerance, accessed by pediatric doctors or parents of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric cardic surgical center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No